CLINICAL TRIAL: NCT06654908
Title: Insulin Resistance and Resisted Exercise Post Burn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Saeed Abd El Aziz Gobara, doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: insulin and resisted exercise
Record Dates: First submitted 2024-10-14; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: (Study group) who have insulin resistance and who will receive resisted exercise (Experimental): This group includes 34 patients who have insulin resistance and who will receive resisted exercise
  Interventions: Procedure: resisted exercise using sand bags,resistance machines and elastic bands
- Group B: (Control group) who have insulin resistance and who will receive routine medical treatment. (No Intervention): This group includes 34 patients who have insulin resistance and who will receive routine medical treatment.

INTERVENTIONS:
Procedure: resisted exercise using sand bags,resistance machines and elastic bands — Rehabilitative exercise training will be performed as previously described. All exercises will be performed using free weights, elastic bands and variable-resistance machines. Modifications to exercises will be made when appropriate depending on the patient injury characteristics. The load will be gradually increased from 50-60% of 3RM at the beginning of the program up to 80-85% of 3RM (repetitions maximum) at the end of the program. All exercise sessions will be preceded by a 5-minute warm-up at <50% VO2peak. No strength training activities will be permitted outside the supervised training session; however, both groups will be encouraged to maintain normal daily activities
  Arms: Group A: (Study group) who have insulin resistance and who will receive resisted exercise

SUMMARY:
The main objective of the present study is to assess the effect of the resisted exercise on insulin resistance post burn.

DETAILED DESCRIPTION:
A burn injury represents the fourth most common type of trauma globally, though it is associated with the most devastating consequences. Severe burn injuries, encompassing 20% of the total body surface area (TBSA) in adults, present a unique challenge compared with other forms of trauma given the magnitude and persistence of systemic deregulation. Indeed, an extensive inflammatory response develops immediately following a severe burn to promote wound healing. This period, known as the "ebb" phase, is comparable with a fight-or-flight response and lasts for the first 72-96 h post injury .

Moreover, burn-induced muscle catabolism places a significant burden on the recovery process, as a 10%-30% loss impairs immune responses and delays wound healing, thereby increasing the risk of infection, and a 40% loss becomes fatal. Despite a mountainous effort to prevent muscle catabolism and wasting. Therefore, a better understanding of the pathophysiology and consequences of burn-induced skeletal muscle wasting is pivotal to alleviating hyper metabolism and reducing morbidity and mortality patients with severe burns .

Hence, extensive burn injury produce clinical syndromes characterized in part by "insulin resistance, it is unclear if these insulin resistant states are identical. To test if the maximal biological effectiveness of insulin is altered in burned patients

ELIGIBILITY:
Inclusion Criteria:

* Patients ranged from 18-35 years of age.
* Patients has waist hip ratio around 0.8 in female and 0.95 in male.
* Patient has body mass index (BMI around 25 kg/m2) (J Obes Weight Loss Ther ,2015).
* Patients has second degree thermal burn injury (superficial and deep partial thickness).
* Patients with around (20% - 40%) of total body surface area (TBSA) burned.
* Patients who are able to follow verbal commands.
* Patients will have upper limb and trunk burn.
* Patients with normal hemoglobin A1C (5.6 %).
* Patients should take diet rich protein, omega 3 and should have good sleep.
* Patients passed two months post severe burns

Exclusion Criteria:

* - Potential participants were excluded if they reported a leg amputation, anoxic brain injury, psychological disorders, quadriplegia, or severe behavior or cognitive disorders history of heart disease, stroke, diabetes mellitus, or any condition that would prevent them from engaging in an exercise study.
* Patients with liver disease, pancreatic disease or any disease affects metabolism.
* If they were already engaging in 2 or more planned exercise sessions per week.
* Patients with any medication to lower glucose levels. Blood pressure and medications to lower lipid levels

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
the outcome of resisted exercises on the improvement of HOMA-IR test results for patients who have around (20% - 40%) of total body surface area (TBSA) burned. | baseline
  sixty-eight patients, who have upper limb and trunk burn. Their ages will be ranged from 18-35 year old. Only patients around (20% - 40%) of total body surface area (TBSA) burned. The participants will be selected from government hospitals (General and insurance hospitals) and randomly distributed into 2 equal groups (group A, group B).
  HOMA-IR analysis measurements:
  All measurements will be taken before the treatment program, 6 weeks after the beginning of treatment program and 12 weeks after the beginning of the treatment program.
  Assessment of insulin resistance:
  • By doing HOMA-IR analysis. HOMA-IR test was performed for both groups before the treatment program, after the 6 weeks of the treatment program and after 12 weeks of the treatment program to evaluate the progression of insulin resistance in both groups.
  The HOMA score of <1.9 was considered as indicator of "Insulin sensitivity"; 1.9 to 2.9 as indicator of "Low IR" and >2.9 as indicator of Significant IR

CONTACTS AND LOCATIONS:
Overall Officials: Amany Rt Abdel Wahid, lecturer, Principal Investigator — Cairo University

REFERENCES:
- [Background] Levy-Marchal C, Arslanian S, Cutfield W, Sinaiko A, Druet C, Marcovecchio ML, Chiarelli F; ESPE-LWPES-ISPAD-APPES-APEG-SLEP-JSPE; Insulin Resistance in Children Consensus Conference Group. Insulin resistance in children: consensus, perspective, and future directions. J Clin Endocrinol Metab. 2010 Dec;95(12):5189-98. doi: 10.1210/jc.2010-1047. Epub 2010 Sep 8. PMID 20829185
- [Background] Angelidi AM, Filippaios A, Mantzoros CS. Severe insulin resistance syndromes. J Clin Invest. 2021 Feb 15;131(4):e142245. doi: 10.1172/JCI142245. PMID 33586681
- [Background] Wallace TM, Matthews DR. The assessment of insulin resistance in man. Diabet Med. 2002 Jul;19(7):527-34. doi: 10.1046/j.1464-5491.2002.00745.x. PMID 12099954
- [Background] Hardee JP, Porter C, Sidossis LS, Borsheim E, Carson JA, Herndon DN, Suman OE. Early rehabilitative exercise training in the recovery from pediatric burn. Med Sci Sports Exerc. 2014 Sep;46(9):1710-6. doi: 10.1249/MSS.0000000000000296. PMID 24824900
- [Background] Lippi G, Ippolito L, Cervellin G. Disseminated intravascular coagulation in burn injury. Semin Thromb Hemost. 2010 Jun;36(4):429-36. doi: 10.1055/s-0030-1254051. Epub 2010 Jul 7. PMID 20614394
- See also: national library of medicine , national centre of biotechnology information — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC11374194/

DOCUMENTS (1):
  • Study Protocol (2024-01-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT06654908/Prot_000.pdf